CLINICAL TRIAL: NCT02676895
Title: A Phase 2a, Observer Blind, Randomized, Controlled, Single Center Study To Evaluate The Safety, Reactogenicity And Immunogenicity Of 2 Doses Of The GVGH 1790GAHB Vaccine Against Shigella Sonnei, Administered Intramuscularly In Adult Subjects From A Country Endemic For Shigellosis
Brief Title: A Study of the Safety and Immune Response of 2 Doses of a New Shigella Vaccine in Kenyan Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205494; H03_04TP (Other: Novartis)
Record Dates: First submitted 2016-02-01; First posted 2016-02-08 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-10

CONDITIONS: Shigella Sonnei Infection
MeSH Terms: interventions — Vaccines; Meningococcal Vaccines; Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1790GAHB 25 μg Group (Experimental): Subjects who received 2 injections of 1790GAHB vaccine containing 25 μg of S. sonnei.
  Interventions: Biological: GVGH S. sonnei (1790GAHB) vaccine 25 μg
- 1790GAHB 100 μg Group (Experimental): Subjects who received 2 injections of 1790GAHB vaccine containing 100 μg of S. sonnei.
  Interventions: Biological: GVGH S. sonnei (1790GAHB) vaccine 100 μg
- Control Group (Active Comparator): Subjects who received one dose of Menveo vaccine and a second dose of Boostrix vaccine.
  Interventions: Biological: Menveo; Biological: Boostrix

INTERVENTIONS:
Biological: GVGH S. sonnei (1790GAHB) vaccine 25 μg — Two injections of the study vaccine were administered 28 days apart.
  Arms: 1790GAHB 25 μg Group
Biological: GVGH S. sonnei (1790GAHB) vaccine 100 μg — Two injections of the study vaccine were administered 28 days apart.
  Arms: 1790GAHB 100 μg Group
Biological: Menveo — One injection of Menveo was administered in subjects in the Control Group.
  Arms: Control Group
Biological: Boostrix — One injection of Boostrix was administered in subjects in the Control Group.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the safety and the immunogenicity of two different doses of the GVGH S. sonnei vaccine in healthy adults and represents the first step towards testing of the GMMA vaccine in the vaccine target population of children from developing countries where shigellosis is endemic.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ≥18 years to ≤45 years of age on the day of informed consent who are resident in the study area and are not planning to leave during the study period.
2. Individuals who, after the nature of the study has been explained, have voluntarily given written consent according to local regulatory requirements, prior to study entry.
3. Individuals who can comply with study procedures including follow-up.
4. Individuals in good health as determined by the outcome of medical history, physical examination, hematology, renal function, and liver function tests, urine dipstick/urinalysis and the clinical judgment of the investigator.
5. Males Or Females of childbearing potential who are using an effective birth control method which they intend to use for the duration of the study Or Females without childbearing potential (i.e. irrespective of birth control method) Prior to receipt of second study vaccination, subjects must be evaluated to confirm that they are eligible for subsequent vaccination. If subjects do not meet any of the original inclusion criteria listed above, they should not receive additional vaccinations.

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
2. Individuals with any progressive or severe neurological disorder, seizure disorder or previous Guillain-Barré syndrome.
3. Individuals who, in the judgment of the investigator, may not be able to comply with all the required study procedures.
4. Individuals with history of any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
5. Individuals with history of reactive arthritis.
6. Individuals with known HIV or hepatitis B virus infection or HIV related disease, history of an autoimmune disorder or any other known or suspected impairment /alteration of the immune system. Individuals under systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 90 days prior to screening.
7. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
8. Individuals with a neutrophil count lower than 1.8 x 10^9/L (applicable to the initial 18 subjects) or lower than 1.0 x 10^9/L (applicable to the additional subjects if approved by DSMB) at screening
9. Individuals with any serious chronic or progressive disease according to judgment of the investigator (e.g., neoplasm, insulin dependent diabetes, Type 2 diabetes mellitus, hypertension, cardiac, renal or hepatic disease and tuberculosis).
10. Individuals who have any malignancy or lymphoproliferative disorder.
11. Individuals with history of allergy to vaccines components or any other allergies deemed by the investigator to increase the risk of an adverse event if they were to participate in the trial.
12. Individuals participating in any clinical trial with another investigational product within 28 days prior to the screening study visit or intent to participate in another clinical study at any time during the conduct of this study.
13. Individuals who received vaccines containing meningococcal A, C, W, Y or tetanus, diphtheria or pertussis antigens within 12 months before screening, or any other vaccines within 4 weeks prior to screening in this study or who are planning to receive any vaccine within the entire study duration.
14. Individuals who have received blood, blood products, and/or plasma derivatives including parenteral immunoglobulin preparations in the 12 weeks prior to the first dose of the study vaccine.
15. Individuals who are study personnel or immediate family members (parents, children, spouse and brothers/sisters) to the personnel conducting this study.
16. Individuals with body temperature > 38.0°C within 3 days of intended study vaccination is a reason for delay of vaccination
17. Individuals with Body Mass Index (BMI)> 30 kg/m^2
18. Individuals with history of substance or alcohol abuse within the past 2 years.
19. Women who are pregnant or are breast-feeding, or are of childbearing age who have not used (for the two months preceding the 1st vaccination) and are not willing to use acceptable contraceptive measures, for the duration of the study. If subjects are women of childbearing potential, they must have a negative pregnancy test at screening visit and prior to enrollment (visit 1). For the purposes of this study acceptable methods of contraception are oral, injected or implantable contraceptives.
20. Individuals who have a previously laboratory confirmed case of disease caused by S. sonnei.
21. Any condition which, in the opinion of the investigator, may pose an increased and unreasonable safety risk to the subject if they participated in the study.
22. Individuals with a previous history of Benign Ethnic Neutropenia or drug related neutropenia.
23. Individuals who have or are likely to require concomitant treatment with neutropenic agents.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 74 enrolled subjects, 2 subjects were allocated numbers but were not administered the study vaccine, hence they did not start the study.
Period: Overall Study
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Started | 22 | 26 | 24
Completed | 20 | 23 | 21
Not Completed | 2 | 3 | 3
Not completed — Administrative reason | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group | Total
Number analyzed (Participants) | 22 | 26 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.6 (5.81) | 26.9 (8.44) | 28.3 (8.23) | 26.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8
  Male | 20 | 23 | 21 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 21 | 26 | 24 | 71
  White | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local and Systemic Adverse Reactions After Each Vaccination
Description: Assessed solicited local adverse reactions were injection site erythema, induration, pain. Assessed systemic adverse reactions were headache, arthralgia, chills, fatigue, malaise, myalgia and temperature (body temperature measured axillary). Any = occurrence of the symptom regardless of intensity grade. Any temperature = body temperature ≥ 38.0°C. Severe symptom = pain, headache, arthralgia, chills, fatigue, malaise and myalgia that prevented normal activity. Severe redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. Severe temperature = body temperature > 40.0 °C.
Time Frame: From 30 minutes up to 7 days following each vaccination
Population: This analysis was performed on the Solicited Safety Set, which included all enrolled subjects who received a study vaccination and for whom solicited adverse event data were available. Less subjects were available to receive the second dose, hence the number or participants analysed is lower for the second dose results.
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 24
Participants
  Any adverse event(s) | 21 | 25 | 21
  Any solicited local adverse event(s) | 21 | 25 | 19
  Any Pain, post-Dose 1 | 20 | 25 | 10
  Severe Pain, post-Dose 1 | 0 | 0 | 0
  Any Erythema, post-Dose 1 | 0 | 0 | 0
  Severe Erythema, post-Dose 1 | 0 | 0 | 0
  Any Induration, post-Dose 1 | 0 | 0 | 0
  Severe Induration, post-Dose 1 | 0 | 0 | 0
  Any Pain, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Pain, post-Dose 2 | 15 | 15 | 17
  Severe Pain, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Pain, post-Dose 2 | 0 | 0 | 0
  Any Erythema, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Erythema, post-Dose 2 | 0 | 0 | 0
  Severe Erythema, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Erythema, post-Dose 2 | 0 | 0 | 0
  Any Induration, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Induration, post-Dose 2 | 0 | 0 | 1
  Severe Induration, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Induration, post-Dose 2 | 0 | 0 | 0
  Any Pain, Across doses | 21 | 25 | 19
  Severe Pain, Across Doses | 0 | 0 | 0
  Any Erythema, Across Doses | 0 | 0 | 0
  Severe Erythema, Across Doses | 0 | 0 | 0
  Any Induration, Across Doses | 0 | 0 | 1
  Severe Induration, Across Doses | 0 | 0 | 0
  Any Solicited systemic adverse event(s) | 9 | 16 | 14
  Any Headache, post-Dose 1 | 5 | 10 | 8
  Severe Headache, post-Dose 1 | 0 | 1 | 0
  Any Arthralgia, post-Dose 1 | 1 | 4 | 4
  Severe Arthralgia, post-Dose 1 | 0 | 0 | 0
  Any Fatigue, post-Dose 1 | 2 | 8 | 7
  Severe Fatigue, post-Dose 1 | 0 | 0 | 0
  Any Chills, post-Dose 1 | 4 | 4 | 3
  Severe Chills, post-Dose 1 | 0 | 0 | 0
  Any Malaise, post-Dose 1 | 3 | 3 | 6
  Severe Malaise, post-Dose 1 | 0 | 0 | 0
  Any Myalgia, post-Dose 1 | 0 | 2 | 2
  Severe Myalgia, post-Dose 1 | 0 | 0 | 0
  Any Temperature, post-Dose 1 | 1 | 1 | 0
  Severe Temperature, post-Dose 1 | 0 | 0 | 0
  Any Headache, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Headache, post-Dose 2 | 4 | 5 | 4
  Severe Headache, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Headache, post-Dose 2 | 0 | 0 | 0
  Any Arthralgia, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Arthralgia, post-Dose 2 | 0 | 0 | 1
  Severe Arthralgia, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Arthralgia, post-Dose 2 | 0 | 0 | 0
  Any Fatigue, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Fatigue, post-Dose 2 | 2 | 1 | 4
  Severe Fatigue, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Fatigue, post-Dose 2 | 0 | 0 | 0
  Any Chills, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Chills, post-Dose 2 | 3 | 1 | 2
  Severe Chills, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Chills, post-Dose 2 | 0 | 0 | 0
  Any Malaise, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Malaise, post-Dose 2 | 2 | 0 | 4
  Severe Malaise, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Malaise, post-Dose 2 | 0 | 0 | 0
  Any Myalgia, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Myalgia, post-Dose 2 | 1 | 0 | 4
  Severe Myalgia, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Myalgia, post-Dose 2 | 0 | 0 | 0
  Any Temperature, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Any Temperature, post-Dose 2 | 0 | 0 | 0
  Severe Temperature, post-Dose 2: number analyzed (Participants) | 22 | 23 | 21
  Severe Temperature, post-Dose 2 | 0 | 0 | 0
  Any Headache, Across Doses | 8 | 13 | 10
  Severe Headache, Across Doses | 0 | 1 | 0
  Any Arthralgia, Across Doses | 1 | 4 | 5
  Severe Arthralgia, Across Doses | 0 | 0 | 0
  Any Fatigue, Across Doses | 3 | 9 | 9
  Severe Fatigue, Across Doses | 0 | 0 | 0
  Any Chills, Across Doses | 5 | 5 | 5
  Severe Chills, Across Doses | 0 | 0 | 0
  Any Malaise, Across Doses | 3 | 3 | 10
  Severe Malaise, Across Doses | 0 | 0 | 0
  Any Myalgia, Across Doses | 1 | 2 | 6
  Severe Myalgia, Across Doses | 0 | 0 | 0
  Any Temperature, Across Doses | 1 | 1 | 0
  Severe Temperature, Across Doses | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is an AE that was not solicited using the Diary Card and that was spontaneously communicated by a subject who has signed the informed consent. Potential unsolicited AEs may be medically attended (defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider), or were of concern to the subject.
  Note: *disruptions= dose reduction, interruption or delay in study vaccination.
Time Frame: During 28 days following each vaccination
Population: This analysis was performed on the Unsolicited Safety Set, which included all enrolled subjects who received a study vaccination and for whom unsolicited adverse event data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 24
Participants
  Any AE | 19 | 24 | 19
  Possibly or Probably related AE | 13 | 16 | 12
  AE leading to study vaccine withdrawal | 0 | 3 | 1
  AE leading to disruptions* | 0 | 3 | 0
  AE leading to hospitalization | 0 | 0 | 0
  AE of special interest (Neutropenia) | 2 | 3 | 1
  Deaths | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that at any dose results in one or more of the following: death; is life-threatening (i.e., the subject was, in the opinion of the investigator, at immediate risk of death from the event as it occurred); it does not refer to an event which hypothetically might have caused death if it were more severe; required or prolonged hospitalization; persistent or significant disability/incapacity (i.e., the event causes a substantial disruption of a person's ability to conduct normal life functions); congenital anomaly/or birth defect; an important and significant medical event that may not be immediately life-threatening or resulting in death or hospitalization but, based upon appropriate medical judgment, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above.
Time Frame: Throughout the whole study period (from Day 1 up to Day 57)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- 1790GAHB 25 μg Group: Subjects who received 2 injections 1790GAHB vaccine containing 25 μg of S. sonnei
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 24
Participants
  Any SAE | 2 | 3 | 1
  Possibly or probably related SAE | 2 | 3 | 1
  Deaths | 0 | 0 | 0

4. Primary Outcome: Number of Subjects With Deviations From Normal Ranges of Safety Laboratory Data at Day 8 by Baseline Ranges
Description: The safety laboratory data included haematological parameters (basophils, eosinophils, erytrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, monocytes, platelets and neutrophils), and chemical parameters (Alkaline Phosphatase [ALP], Alanine Aminotransferase [ALA], Aspartate Aminotransferase [AST], Bilirubin [BILI], Blood Urea Nitrogen [BUN], Creatinine [CREAT], Gamma Glutamyl Transferase [GGT], Glucose [GLUC], Potassium [K], Lactate Dehydrogenase [LDH] and Sodium [Na]).
  Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 8 (7 days after first vaccination)
Population: This analysis was performed on the Overall Safety Set, which included all enrolled subjects who received a study vaccination and for whom solicited and/or unsolicited adverse event data were available. Less subjects were available with each subsequent visit, hence the number of subjects analysed is lower than in the previous timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 23
Participants
  Basophils: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 8) | 9 | 9 | 5
  Basophils: Above (baseline) - within (Day 8) | 3 | 5 | 6
  Basophils: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 8) | 3 | 1 | 2
  Basophils: Above (baseline) - above (Day 8) | 7 | 11 | 10
  Eosinophils: Below (baseline) - below (Day 8) | 0 | 0 | 1
  Eosinophils: Within (baseline) - below (Day 8) | 1 | 1 | 0
  Eosinophils: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 8) | 1 | 1 | 0
  Eosinophils: Within (baseline) - within (Day 8) | 20 | 24 | 22
  Eosinophils: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Erythrocytes: Below (baseline) - below (Day 8) | 0 | 0 | 1
  Erythrocytes: Within (baseline) - below (Day 8) | 1 | 0 | 0
  Erythrocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Erythrocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Erythrocytes: Within (baseline) - within (Day 8) | 20 | 24 | 22
  Erythrocytes: Above (baseline) - within (Day 8) | 0 | 2 | 0
  Erythrocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Erythrocytes: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Erythrocytes: Above (baseline) - above (Day 8) | 1 | 0 | 0
  Hematocrit: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Hematocrit: Within (baseline) - below (Day 8) | 0 | 1 | 0
  Hematocrit: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Hematocrit: Below (baseline) - within (Day 8) | 0 | 0 | 1
  Hematocrit: Within (baseline) - within (Day 8) | 22 | 21 | 22
  Hematocrit: Above (baseline) - within (Day 8) | 0 | 3 | 0
  Hematocrit: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Hematocrit: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Hematocrit: Above (baseline) - above (Day 8) | 0 | 1 | 0
  Hemoglobin: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 8) | 0 | 1 | 0
  Hemoglobin: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 8) | 22 | 24 | 23
  Hemoglobin: Above (baseline) - within (Day 8) | 0 | 1 | 0
  Hemoglobin: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Leukocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Leukocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Leukocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Leukocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Leukocytes: Within (baseline) - within (Day 8) | 21 | 25 | 22
  Leukocytes: Above (baseline) - within (Day 8) | 1 | 1 | 0
  Leukocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Leukocytes: Within (baseline) - above (Day 8) | 0 | 0 | 1
  Leukocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 8) | 2 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 8) | 19 | 26 | 22
  Lymphocytes: Above (baseline) - within (Day 8) | 1 | 0 | 1
  Lymphocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 8) | 2 | 2 | 4
  Monocytes: Within (baseline) - below (Day 8) | 2 | 2 | 3
  Monocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 8) | 3 | 7 | 3
  Monocytes: Within (baseline) - within (Day 8) | 15 | 15 | 13
  Monocytes: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Monocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 8) | 22 | 26 | 22
  Neutrophils: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Neutrophils: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 8) | 0 | 0 | 1
  Neutrophils: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Platelets: Below (baseline) - below (Day 8) | 0 | 3 | 0
  Platelets: Within (baseline) - below (Day 8) | 2 | 0 | 2
  Platelets: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Platelets: Within (baseline) - within (Day 8) | 19 | 21 | 21
  Platelets: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Platelets: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 8) | 0 | 2 | 0
  Platelets: Above (baseline) - above (Day 8) | 1 | 0 | 0
  ALA: Below (baseline) - below (Day 8) | 0 | 0 | 0
  ALA: Within (baseline) - below (Day 8) | 0 | 0 | 0
  ALA: Above (baseline) - below (Day 8) | 0 | 0 | 0
  ALA: Below (baseline) - within (Day 8) | 0 | 0 | 0
  ALA: Within (baseline) - within (Day 8) | 22 | 26 | 23
  ALA: Above (baseline) - within (Day 8) | 0 | 0 | 0
  ALA: Below (baseline) - above (Day 8) | 0 | 0 | 0
  ALA: Within (baseline) - above (Day 8) | 0 | 0 | 0
  ALA: Above (baseline) - above (Day 8) | 0 | 0 | 0
  ALP: Below (baseline) - below (Day 8) | 0 | 0 | 0
  ALP: Within (baseline) - below (Day 8) | 0 | 0 | 0
  ALP: Above (baseline) - below (Day 8) | 0 | 0 | 0
  ALP: Below (baseline) - within (Day 8) | 0 | 0 | 0
  ALP: Within (baseline) - within (Day 8) | 21 | 25 | 21
  ALP: Above (baseline) - within (Day 8) | 1 | 0 | 1
  ALP: Below (baseline) - above (Day 8) | 0 | 0 | 0
  ALP: Within (baseline) - above (Day 8) | 0 | 0 | 1
  ALP: Above (baseline) - above (Day 8) | 0 | 1 | 0
  AST: Below (baseline) - below (Day 8) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 8) | 0 | 1 | 0
  AST: Above (baseline) - below (Day 8) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 8) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 8) | 22 | 23 | 23
  AST: Above (baseline) - within (Day 8) | 0 | 2 | 0
  AST: Below (baseline) - above (Day 8) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 8) | 0 | 0 | 0
  AST: Above (baseline) - above (Day 8) | 0 | 0 | 0
  BILI: Below (baseline) - below (Day 8) | 1 | 0 | 0
  BILI: Within (baseline) - below (Day 8) | 2 | 1 | 2
  BILI: Above (baseline) - below (Day 8) | 0 | 0 | 0
  BILI: Below (baseline) - within (Day 8) | 2 | 1 | 1
  BILI: Within (baseline) - within (Day 8) | 17 | 22 | 20
  BILI: Above (baseline) - within (Day 8) | 0 | 1 | 0
  BILI: Below (baseline) - above (Day 8) | 0 | 0 | 0
  BILI: Within (baseline) - above (Day 8) | 0 | 1 | 0
  BILI: Above (baseline) - above (Day 8) | 0 | 0 | 0
  BUN: Below (baseline) - below (Day 8) | 0 | 0 | 0
  BUN: Within (baseline) - below (Day 8) | 1 | 7 | 0
  BUN: Above (baseline) - below (Day 8) | 0 | 0 | 0
  BUN: Below (baseline) - within (Day 8) | 1 | 1 | 1
  BUN: Within (baseline) - within (Day 8) | 20 | 18 | 22
  BUN: Above (baseline) - within (Day 8) | 0 | 0 | 0
  BUN: Below (baseline) - above (Day 8) | 0 | 0 | 0
  BUN: Within (baseline) - above (Day 8) | 0 | 0 | 0
  BUN: Above (baseline) - above (Day 8) | 0 | 0 | 0
  CREA: Below (baseline) - below (Day 8) | 0 | 0 | 0
  CREA: Within (baseline) - below (Day 8) | 0 | 1 | 0
  CREA: Above (baseline) - below (Day 8) | 0 | 0 | 0
  CREA: Below (baseline) - within (Day 8) | 0 | 0 | 0
  CREA: Within (baseline) - within (Day 8) | 20 | 23 | 19
  CREA: Above (baseline) - within (Day 8) | 1 | 0 | 1
  CREA: Below (baseline) - above (Day 8) | 0 | 0 | 0
  CREA: Within (baseline) - above (Day 8) | 1 | 1 | 3
  CREA: Above (baseline) - above (Day 8) | 0 | 1 | 0
  GGT: Below (baseline) - below (Day 8) | 0 | 0 | 0
  GGT: Within (baseline) - below (Day 8) | 0 | 0 | 0
  GGT: Above (baseline) - below (Day 8) | 0 | 0 | 0
  GGT: Below (baseline) - within (Day 8) | 0 | 0 | 0
  GGT: Within (baseline) - within (Day 8) | 21 | 23 | 20
  GGT: Above (baseline) - within (Day 8) | 1 | 0 | 1
  GGT: Below (baseline) - above (Day 8) | 0 | 0 | 0
  GGT: Within (baseline) - above (Day 8) | 0 | 0 | 0
  GGT: Above (baseline) - above (Day 8) | 0 | 3 | 2
  GLUC: Below (baseline) - below (Day 8) | 0 | 0 | 0
  GLUC: Within (baseline) - below (Day 8) | 1 | 0 | 0
  GLUC: Above (baseline) - below (Day 8) | 0 | 0 | 0
  GLUC: Below (baseline) - within (Day 8) | 0 | 0 | 0
  GLUC: Within (baseline) - within (Day 8) | 21 | 26 | 21
  GLUC: Above (baseline) - within (Day 8) | 0 | 0 | 0
  GLUC: Below (baseline) - above (Day 8) | 0 | 0 | 0
  GLUC: Within (baseline) - above (Day 8) | 0 | 0 | 2
  GLUC: Above (baseline) - above (Day 8) | 0 | 0 | 0
  LDH: Below (baseline) - below (Day 8) | 0 | 0 | 0
  LDH: Within (baseline) - below (Day 8) | 1 | 0 | 1
  LDH: Above (baseline) - below (Day 8) | 0 | 0 | 0
  LDH: Below (baseline) - within (Day 8) | 0 | 0 | 0
  LDH: Within (baseline) - within (Day 8) | 21 | 26 | 22
  LDH: Above (baseline) - within (Day 8) | 0 | 0 | 0
  LDH: Below (baseline) - above (Day 8) | 0 | 0 | 0
  LDH: Within (baseline) - above (Day 8) | 0 | 0 | 0
  LDH: Above (baseline) - above (Day 8) | 0 | 0 | 0
  K: Below (baseline) - below (Day 8) | 0 | 0 | 0
  K: Within (baseline) - below (Day 8) | 0 | 0 | 0
  K: Above (baseline) - below (Day 8) | 0 | 0 | 0
  K: Below (baseline) - within (Day 8) | 0 | 0 | 0
  K: Within (baseline) - within (Day 8) | 15 | 16 | 19
  K: Above (baseline) - within (Day 8) | 2 | 2 | 3
  K: Below (baseline) - above (Day 8) | 0 | 0 | 0
  K: Within (baseline) - above (Day 8) | 4 | 6 | 1
  K: Above (baseline) - above (Day 8) | 1 | 2 | 0
  Na: Below (baseline) - below (Day 8) | 0 | 1 | 0
  Na: Within (baseline) - below (Day 8) | 1 | 2 | 2
  Na: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Na: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Na: Within (baseline) - within (Day 8) | 21 | 23 | 21
  Na: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Na: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Na: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Na: Above (baseline) - above (Day 8) | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Deviations From Normal Ranges of Safety Laboratory Data at Day 29 by Baseline Ranges
Description: as for outcome 4
Time Frame: At Day 29 (28 days after the first vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 22
Participants
  Basophils: number analyzed (Participants) | 21 | 26 | 22
  Basophils: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 29) | 9 | 8 | 4
  Basophils: Above (baseline) - within (Day 29) | 4 | 4 | 7
  Basophils: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 29) | 2 | 2 | 3
  Basophils: Above (baseline) - above (Day 29) | 6 | 12 | 8
  Eosinophils: number analyzed (Participants) | 21 | 26 | 22
  Eosinophils: Below (baseline) - below (Day 29) | 0 | 0 | 1
  Eosinophils: Within (baseline) - below (Day 29) | 0 | 1 | 0
  Eosinophils: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 29) | 1 | 1 | 0
  Eosinophils: Within (baseline) - within (Day 29) | 20 | 24 | 20
  Eosinophils: Above (baseline) - within (Day 29) | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 29) | 0 | 0 | 1
  Eosinophils: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Erythrocytes: number analyzed (Participants) | 21 | 26 | 22
  Erythrocytes: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Erythrocytes: Within (baseline) - below (Day 29) | 1 | 0 | 0
  Erythrocytes: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Erythrocytes: Below (baseline) - within (Day 29) | 0 | 0 | 1
  Erythrocytes: Within (baseline) - within (Day 29) | 19 | 24 | 21
  Erythrocytes: Above (baseline) - within (Day 29) | 0 | 1 | 0
  Erythrocytes: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Erythrocytes: Within (baseline) - above (Day 29) | 0 | 0 | 0
  Erythrocytes: Above (baseline) - above (Day 29) | 1 | 1 | 0
  Hematocrit: number analyzed (Participants) | 21 | 26 | 22
  Hematocrit: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Hematocrit: Within (baseline) - below (Day 29) | 0 | 1 | 0
  Hematocrit: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Hematocrit: Below (baseline) - within (Day 29) | 0 | 0 | 1
  Hematocrit: Within (baseline) - within (Day 29) | 21 | 21 | 21
  Hematocrit: Above (baseline) - within (Day 29) | 0 | 4 | 0
  Hematocrit: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Hematocrit: Within (baseline) - above (Day 29) | 0 | 0 | 0
  Hematocrit: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Hemoglobin: number analyzed (Participants) | 21 | 26 | 22
  Hemoglobin: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 29) | 0 | 1 | 0
  Hemoglobin: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 29) | 21 | 24 | 22
  Hemoglobin: Above (baseline) - within (Day 29) | 0 | 1 | 0
  Hemoglobin: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 29) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Leukocytes: number analyzed (Participants) | 21 | 26 | 22
  Leukocytes: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Leukocytes: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Leukocytes: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Leukocytes: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Leukocytes: Within (baseline) - within (Day 29) | 20 | 24 | 22
  Leukocytes: Above (baseline) - within (Day 29) | 1 | 1 | 0
  Leukocytes: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Leukocytes: Within (baseline) - above (Day 29) | 0 | 1 | 0
  Leukocytes: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Lymphocytes: number analyzed (Participants) | 21 | 26 | 22
  Lymphocytes: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 29) | 20 | 24 | 21
  Lymphocytes: Above (baseline) - within (Day 29) | 1 | 0 | 1
  Lymphocytes: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 29) | 0 | 2 | 0
  Lymphocytes: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Monocytes: number analyzed (Participants) | 21 | 26 | 22
  Monocytes: Below (baseline) - below (Day 29) | 3 | 4 | 1
  Monocytes: Within (baseline) - below (Day 29) | 1 | 1 | 1
  Monocytes: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 29) | 2 | 5 | 6
  Monocytes: Within (baseline) - within (Day 29) | 15 | 15 | 14
  Monocytes: Above (baseline) - within (Day 29) | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 29) | 0 | 1 | 0
  Monocytes: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Neutrophils: number analyzed (Participants) | 21 | 26 | 22
  Neutrophils: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 29) | 21 | 25 | 22
  Neutrophils: Above (baseline) - within (Day 29) | 0 | 0 | 0
  Neutrophils: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 29) | 0 | 1 | 0
  Neutrophils: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Platelets: number analyzed (Participants) | 21 | 26 | 22
  Platelets: Below (baseline) - below (Day 29) | 0 | 2 | 0
  Platelets: Within (baseline) - below (Day 29) | 1 | 0 | 2
  Platelets: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 29) | 0 | 1 | 0
  Platelets: Within (baseline) - within (Day 29) | 19 | 22 | 20
  Platelets: Above (baseline) - within (Day 29) | 1 | 0 | 0
  Platelets: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 29) | 0 | 1 | 0
  Platelets: Above (baseline) - above (Day 29) | 0 | 0 | 0
  ALA: Below (baseline) - below (Day 29) | 0 | 0 | 0
  ALA: Within (baseline) - below (Day 29) | 0 | 0 | 0
  ALA: Above (baseline) - below (Day 29) | 0 | 0 | 0
  ALA: Below (baseline) - within (Day 29) | 0 | 0 | 0
  ALA: Within (baseline) - within (Day 29) | 22 | 26 | 22
  ALA: Above (baseline) - within (Day 29) | 0 | 0 | 0
  ALA: Below (baseline) - above (Day 29) | 0 | 0 | 0
  ALA: Within (baseline) - above (Day 29) | 0 | 0 | 0
  ALA: Above (baseline) - above (Day 29) | 0 | 0 | 0
  ALP: Below (baseline) - below (Day 29) | 0 | 0 | 0
  ALP: Within (baseline) - below (Day 29) | 0 | 2 | 1
  ALP: Above (baseline) - below (Day 29) | 0 | 0 | 0
  ALP: Below (baseline) - within (Day 29) | 0 | 0 | 0
  ALP: Within (baseline) - within (Day 29) | 21 | 23 | 19
  ALP: Above (baseline) - within (Day 29) | 1 | 1 | 0
  ALP: Below (baseline) - above (Day 29) | 0 | 0 | 0
  ALP: Within (baseline) - above (Day 29) | 0 | 0 | 1
  ALP: Above (baseline) - above (Day 29) | 0 | 0 | 1
  AST: Below (baseline) - below (Day 29) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 29) | 1 | 1 | 0
  AST: Above (baseline) - below (Day 29) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 29) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 29) | 21 | 22 | 22
  AST: Above (baseline) - within (Day 29) | 0 | 1 | 0
  AST: Below (baseline) - above (Day 29) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 29) | 0 | 1 | 0
  AST: Above (baseline) - above (Day 29) | 0 | 1 | 0
  BILI: Below (baseline) - below (Day 29) | 1 | 0 | 0
  BILI: Within (baseline) - below (Day 29) | 0 | 1 | 0
  BILI: Above (baseline) - below (Day 29) | 0 | 0 | 0
  BILI: Below (baseline) - within (Day 29) | 2 | 1 | 1
  BILI: Within (baseline) - within (Day 29) | 19 | 23 | 21
  BILI: Above (baseline) - within (Day 29) | 0 | 1 | 0
  BILI: Below (baseline) - above (Day 29) | 0 | 0 | 0
  BILI: Within (baseline) - above (Day 29) | 0 | 0 | 0
  BILI: Above (baseline) - above (Day 29) | 0 | 0 | 0
  BUN: Below (baseline) - below (Day 29) | 0 | 0 | 0
  BUN: Within (baseline) - below (Day 29) | 1 | 1 | 0
  BUN: Above (baseline) - below (Day 29) | 0 | 0 | 0
  BUN: Below (baseline) - within (Day 29) | 1 | 1 | 1
  BUN: Within (baseline) - within (Day 29) | 20 | 24 | 21
  BUN: Above (baseline) - within (Day 29) | 0 | 0 | 0
  BUN: Below (baseline) - above (Day 29) | 0 | 0 | 0
  BUN: Within (baseline) - above (Day 29) | 0 | 0 | 0
  BUN: Above (baseline) - above (Day 29) | 0 | 0 | 0
  CREA: Below (baseline) - below (Day 29) | 0 | 0 | 0
  CREA: Within (baseline) - below (Day 29) | 0 | 0 | 0
  CREA: Above (baseline) - below (Day 29) | 0 | 0 | 0
  CREA: Below (baseline) - within (Day 29) | 0 | 0 | 0
  CREA: Within (baseline) - within (Day 29) | 21 | 22 | 19
  CREA: Above (baseline) - within (Day 29) | 0 | 0 | 1
  CREA: Below (baseline) - above (Day 29) | 0 | 0 | 0
  CREA: Within (baseline) - above (Day 29) | 0 | 3 | 2
  CREA: Above (baseline) - above (Day 29) | 1 | 1 | 0
  GGT: Below (baseline) - below (Day 29) | 0 | 0 | 0
  GGT: Within (baseline) - below (Day 29) | 0 | 0 | 0
  GGT: Above (baseline) - below (Day 29) | 0 | 0 | 0
  GGT: Below (baseline) - within (Day 29) | 0 | 0 | 0
  GGT: Within (baseline) - within (Day 29) | 18 | 21 | 18
  GGT: Above (baseline) - within (Day 29) | 1 | 0 | 1
  GGT: Below (baseline) - above (Day 29) | 0 | 0 | 0
  GGT: Within (baseline) - above (Day 29) | 3 | 2 | 1
  GGT: Above (baseline) - above (Day 29) | 0 | 3 | 2
  GLUC: Below (baseline) - below (Day 29) | 0 | 0 | 0
  GLUC: Within (baseline) - below (Day 29) | 0 | 0 | 0
  GLUC: Above (baseline) - below (Day 29) | 0 | 0 | 0
  GLUC: Below (baseline) - within (Day 29) | 0 | 0 | 0
  GLUC: Within (baseline) - within (Day 29) | 22 | 26 | 21
  GLUC: Above (baseline) - within (Day 29) | 0 | 0 | 0
  GLUC: Below (baseline) - above (Day 29) | 0 | 0 | 0
  GLUC: Within (baseline) - above (Day 29) | 0 | 0 | 1
  GLUC: Above (baseline) - above (Day 29) | 0 | 0 | 0
  LDH: Below (baseline) - below (Day 29) | 0 | 0 | 0
  LDH: Within (baseline) - below (Day 29) | 0 | 1 | 1
  LDH: Above (baseline) - below (Day 29) | 0 | 0 | 0
  LDH: Below (baseline) - within (Day 29) | 0 | 0 | 0
  LDH: Within (baseline) - within (Day 29) | 21 | 23 | 19
  LDH: Above (baseline) - within (Day 29) | 0 | 0 | 0
  LDH: Below (baseline) - above (Day 29) | 0 | 0 | 0
  LDH: Within (baseline) - above (Day 29) | 1 | 2 | 2
  LDH: Above (baseline) - above (Day 29) | 0 | 0 | 0
  K: Below (baseline) - below (Day 29) | 0 | 0 | 0
  K: Within (baseline) - below (Day 29) | 0 | 1 | 0
  K: Above (baseline) - below (Day 29) | 0 | 0 | 0
  K: Below (baseline) - within (Day 29) | 0 | 0 | 0
  K: Within (baseline) - within (Day 29) | 19 | 15 | 16
  K: Above (baseline) - within (Day 29) | 1 | 4 | 2
  K: Below (baseline) - above (Day 29) | 0 | 0 | 0
  K: Within (baseline) - above (Day 29) | 0 | 6 | 4
  K: Above (baseline) - above (Day 29) | 2 | 0 | 0
  Na: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Na: Within (baseline) - below (Day 29) | 4 | 6 | 2
  Na: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Na: Below (baseline) - within (Day 29) | 0 | 1 | 0
  Na: Within (baseline) - within (Day 29) | 18 | 19 | 20
  Na: Above (baseline) - within (Day 29) | 0 | 0 | 0
  Na: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Na: Within (baseline) - above (Day 29) | 0 | 0 | 0
  Na: Above (baseline) - above (Day 29) | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Deviations From Normal Ranges of Safety Laboratory Data at Day 36 by Baseline Ranges
Description: as for outcome 4
Time Frame: At Day 36 (7 days after the second vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 24 | 21
Participants
  Basophils: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 36) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Basophils: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 36) | 9 | 7 | 5
  Basophils: Above (baseline) - within (Day 36) | 2 | 6 | 5
  Basophils: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 36) | 3 | 1 | 2
  Basophils: Above (baseline) - above (Day 36) | 8 | 10 | 9
  Eosinophils: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 36) | 0 | 1 | 1
  Eosinophils: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Eosinophils: Below (baseline) - Within (Day 36) | 1 | 1 | 1
  Eosinophils: Within (baseline) - within (Day 36) | 21 | 22 | 18
  Eosinophils: Above (baseline) - within (Day 36) | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 36) | 0 | 0 | 1
  Eosinophils: Above (baseline) - above (Day 36) | 0 | 0 | 0
  Erythrocytes: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Erythrocytes: Within (baseline) - below (Day 36) | 1 | 0 | 0
  Erythrocytes: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Erythrocytes: Below (baseline) - Within (Day 36) | 0 | 0 | 1
  Erythrocytes: Within (baseline) - within (Day 36) | 20 | 22 | 20
  Erythrocytes: Above (baseline) - within (Day 36) | 0 | 1 | 0
  Erythrocytes: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Erythrocytes: Within (baseline) - above (Day 36) | 0 | 0 | 0
  Erythrocytes: Above (baseline) - above (Day 36) | 1 | 1 | 0
  Hematocrit: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Hematocrit: Within (baseline) - below (Day 36) | 0 | 0 | 0
  Hematocrit: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Hematocrit: Below (baseline) - Within (Day 36) | 0 | 0 | 1
  Hematocrit: Within (baseline) - within (Day 36) | 22 | 20 | 20
  Hematocrit: Above (baseline) - within (Day 36) | 0 | 4 | 0
  Hematocrit: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Hematocrit: Within (baseline) - above (Day 36) | 0 | 0 | 0
  Hematocrit: Above (baseline) - above (Day 36) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 36) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 36) | 22 | 23 | 21
  Hemoglobin: Above (baseline) - within (Day 36) | 0 | 1 | 0
  Hemoglobin: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 36) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 36) | 0 | 0 | 0
  Leukocytes: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Leukocytes: Within (baseline) - below (Day 36) | 0 | 0 | 0
  Leukocytes: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Leukocytes: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  Leukocytes: Within (baseline) - within (Day 36) | 21 | 22 | 21
  Leukocytes: Above (baseline) - within (Day 36) | 1 | 1 | 0
  Leukocytes: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Leukocytes: Within (baseline) - above (Day 36) | 0 | 1 | 0
  Leukocytes: Above (baseline) - above (Day 36) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 36) | 1 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 36) | 20 | 23 | 19
  Lymphocytes: Above (baseline) - within (Day 36) | 1 | 0 | 1
  Lymphocytes: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 36) | 0 | 1 | 1
  Lymphocytes: Above (baseline) - above (Day 36) | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 36) | 1 | 2 | 3
  Monocytes: Within (baseline) - below (Day 36) | 2 | 0 | 3
  Monocytes: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Monocytes: Below (baseline) - Within (Day 36) | 4 | 6 | 4
  Monocytes: Within (baseline) - within (Day 36) | 15 | 15 | 11
  Monocytes: Above (baseline) - within (Day 36) | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 36) | 0 | 1 | 0
  Monocytes: Above (baseline) - above (Day 36) | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 36) | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Neutrophils: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 36) | 22 | 24 | 21
  Neutrophils: Above (baseline) - within (Day 36) | 0 | 0 | 0
  Neutrophils: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 36) | 0 | 0 | 0
  Neutrophils: Above (baseline) - above (Day 36) | 0 | 0 | 0
  Platelet: Below (baseline) - below (Day 36) | 0 | 2 | 0
  Platelet: Within (baseline) - below (Day 36) | 1 | 0 | 2
  Platelet: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Platelet: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  Platelet: Within (baseline) - within (Day 36) | 20 | 22 | 19
  Platelet: Above (baseline) - within (Day 36) | 0 | 0 | 0
  Platelet: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Platelet: Within (baseline) - above (Day 36) | 0 | 0 | 0
  Platelet: Above (baseline) - above (Day 36) | 1 | 0 | 0
  ALA: Below (baseline) - below (Day 36) | 0 | 0 | 0
  ALA: Within (baseline) - below (Day 36) | 0 | 0 | 0
  ALA: Above (baseline) - below (Day 36) | 0 | 0 | 0
  ALA: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  ALA: Within (baseline) - within (Day 36) | 22 | 24 | 21
  ALA: Above (baseline) - within (Day 36) | 0 | 0 | 0
  ALA: Below (baseline) - above (Day 36) | 0 | 0 | 0
  ALA: Within (baseline) - above (Day 36) | 0 | 0 | 0
  ALA: Above (baseline) - above (Day 36) | 0 | 0 | 0
  ALP: Below (baseline) - below (Day 36) | 0 | 0 | 0
  ALP: Within (baseline) - below (Day 36) | 0 | 0 | 1
  ALP: Above (baseline) - below (Day 36) | 0 | 0 | 0
  ALP: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  ALP: Within (baseline) - within (Day 36) | 20 | 22 | 19
  ALP: Above (baseline) - within (Day 36) | 1 | 0 | 0
  ALP: Below (baseline) - above (Day 36) | 0 | 0 | 0
  ALP: Within (baseline) - above (Day 36) | 1 | 1 | 0
  ALP: Above (baseline) - above (Day 36) | 0 | 1 | 1
  AST: Below (baseline) - below (Day 36) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 36) | 1 | 1 | 0
  AST: Above (baseline) - below (Day 36) | 0 | 0 | 0
  AST: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 36) | 20 | 21 | 20
  AST: Above (baseline) - within (Day 36) | 0 | 1 | 0
  AST: Below (baseline) - above (Day 36) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 36) | 1 | 0 | 1
  AST: Above (baseline) - above (Day 36) | 0 | 1 | 0
  BILI: Below (baseline) - below (Day 36) | 0 | 0 | 0
  BILI: Within (baseline) - below (Day 36) | 3 | 1 | 0
  BILI: Above (baseline) - below (Day 36) | 0 | 0 | 0
  BILI: Below (baseline) - Within (Day 36) | 3 | 1 | 1
  BILI: Within (baseline) - within (Day 36) | 16 | 21 | 20
  BILI: Above (baseline) - within (Day 36) | 0 | 1 | 0
  BILI: Below (baseline) - above (Day 36) | 0 | 0 | 0
  BILI: Within (baseline) - above (Day 36) | 0 | 0 | 0
  BILI: Above (baseline) - above (Day 36) | 0 | 0 | 0
  BUN: Below (baseline) - below (Day 36) | 0 | 1 | 0
  BUN: Within (baseline) - below (Day 36) | 2 | 0 | 0
  BUN: Above (baseline) - below (Day 36) | 0 | 0 | 0
  BUN: Below (baseline) - Within (Day 36) | 1 | 0 | 1
  BUN: Within (baseline) - within (Day 36) | 19 | 23 | 20
  BUN: Above (baseline) - within (Day 36) | 0 | 0 | 0
  BUN: Below (baseline) - above (Day 36) | 0 | 0 | 0
  BUN: Within (baseline) - above (Day 36) | 0 | 0 | 0
  BUN: Above (baseline) - above (Day 36) | 0 | 0 | 0
  CREA: Below (baseline) - below (Day 36) | 0 | 0 | 0
  CREA: Within (baseline) - below (Day 36) | 0 | 1 | 0
  CREA: Above (baseline) - below (Day 36) | 0 | 0 | 0
  CREA: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  CREA: Within (baseline) - within (Day 36) | 20 | 17 | 18
  CREA: Above (baseline) - within (Day 36) | 1 | 1 | 0
  CREA: Below (baseline) - above (Day 36) | 0 | 0 | 0
  CREA: Within (baseline) - above (Day 36) | 1 | 5 | 2
  CREA: Above (baseline) - above (Day 36) | 0 | 0 | 1
  GGT: Below (baseline) - below (Day 36) | 0 | 0 | 0
  GGT: Within (baseline) - below (Day 36) | 0 | 0 | 0
  GGT: Above (baseline) - below (Day 36) | 0 | 0 | 0
  GGT: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  GGT: Within (baseline) - within (Day 36) | 19 | 19 | 18
  GGT: Above (baseline) - within (Day 36) | 0 | 2 | 1
  GGT: Below (baseline) - above (Day 36) | 0 | 0 | 0
  GGT: Within (baseline) - above (Day 36) | 2 | 3 | 1
  GGT: Above (baseline) - above (Day 36) | 1 | 0 | 1
  GLUC: Below (baseline) - below (Day 36) | 0 | 0 | 0
  GLUC: Within (baseline) - below (Day 36) | 0 | 0 | 0
  GLUC: Above (baseline) - below (Day 36) | 0 | 0 | 0
  GLUC: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  GLUC: Within (baseline) - within (Day 36) | 22 | 24 | 21
  GLUC: Above (baseline) - within (Day 36) | 0 | 0 | 0
  GLUC: Below (baseline) - above (Day 36) | 0 | 0 | 0
  GLUC: Within (baseline) - above (Day 36) | 0 | 0 | 0
  GLUC: Above (baseline) - above (Day 36) | 0 | 0 | 0
  LDH: Below (baseline) - below (Day 36) | 0 | 0 | 0
  LDH: Within (baseline) - below (Day 36) | 1 | 0 | 1
  LDH: Above (baseline) - below (Day 36) | 0 | 0 | 0
  LDH: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  LDH: Within (baseline) - within (Day 36) | 20 | 23 | 19
  LDH: Above (baseline) - within (Day 36) | 0 | 0 | 0
  LDH: Below (baseline) - above (Day 36) | 0 | 0 | 0
  LDH: Within (baseline) - above (Day 36) | 1 | 1 | 1
  LDH: Above (baseline) - above (Day 36) | 0 | 0 | 0
  K: Below (baseline) - below (Day 36) | 0 | 0 | 0
  K: Within (baseline) - below (Day 36) | 0 | 0 | 1
  K: Above (baseline) - below (Day 36) | 0 | 0 | 0
  K: Below (baseline) - Within (Day 36) | 0 | 0 | 0
  K: Within (baseline) - within (Day 36) | 8 | 13 | 15
  K: Above (baseline) - within (Day 36) | 2 | 4 | 2
  K: Below (baseline) - above (Day 36) | 0 | 0 | 0
  K: Within (baseline) - above (Day 36) | 11 | 7 | 3
  K: Above (baseline) - above (Day 36) | 1 | 0 | 0
  Na: Below (baseline) - below (Day 36) | 0 | 0 | 0
  Na: Within (baseline) - below (Day 36) | 1 | 2 | 0
  Na: Above (baseline) - below (Day 36) | 0 | 0 | 0
  Na: Below (baseline) - Within (Day 36) | 0 | 1 | 0
  Na: Within (baseline) - within (Day 36) | 21 | 20 | 21
  Na: Above (baseline) - within (Day 36) | 0 | 0 | 0
  Na: Below (baseline) - above (Day 36) | 0 | 0 | 0
  Na: Within (baseline) - above (Day 36) | 0 | 1 | 0
  Na: Above (baseline) - above (Day 36) | 0 | 0 | 0

7. Primary Outcome: Number of Subjects With Deviations From Normal Ranges of Safety Laboratory Data at Day 57 by Baseline Ranges
Description: as for outcome 4
Time Frame: At Day 57 (28 days after the second vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 21 | 23 | 21
Participants
  Basophils: Below (baseline) - below (Day 57) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 57) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 57) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 57) | 8 | 7 | 6
  Basophils: Above (baseline) - within (Day 57) | 5 | 7 | 8
  Basophils: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 57) | 4 | 1 | 1
  Basophils: Above (baseline) - above (Day 57) | 4 | 8 | 6
  Eosinophils: Below (baseline) - below (Day 57) | 0 | 1 | 0
  Eosinophils: Within (baseline) - below (Day 57) | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 57) | 1 | 0 | 1
  Eosinophils: Within (baseline) - within (Day 57) | 20 | 22 | 18
  Eosinophils: Above (baseline) - within (Day 57) | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 57) | 0 | 0 | 2
  Eosinophils: Above (baseline) - above (Day 57) | 0 | 0 | 0
  Erythrocytes: Below (baseline) - below (Day 57) | 0 | 0 | 0
  Erythrocytes: Within (baseline) - below (Day 57) | 0 | 0 | 0
  Erythrocytes: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Erythrocytes: Below (baseline) - within (Day 57) | 0 | 0 | 1
  Erythrocytes: Within (baseline) - within (Day 57) | 20 | 21 | 20
  Erythrocytes: Above (baseline) - within (Day 57) | 0 | 2 | 0
  Erythrocytes: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Erythrocytes: Within (baseline) - above (Day 57) | 0 | 0 | 0
  Erythrocytes: Above (baseline) - above (Day 57) | 1 | 0 | 0
  Hematocrit: Below (baseline) - below (Day 57) | 0 | 0 | 0
  Hematocrit: Within (baseline) - below (Day 57) | 1 | 0 | 0
  Hematocrit: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Hematocrit: Below (baseline) - within (Day 57) | 0 | 0 | 1
  Hematocrit: Within (baseline) - within (Day 57) | 20 | 20 | 20
  Hematocrit: Above (baseline) - within (Day 57) | 0 | 3 | 0
  Hematocrit: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Hematocrit: Within (baseline) - above (Day 57) | 0 | 0 | 0
  Hematocrit: Above (baseline) - above (Day 57) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 57) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 57) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 57) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 57) | 21 | 22 | 21
  Hemoglobin: Above (baseline) - within (Day 57) | 0 | 1 | 0
  Hemoglobin: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 57) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 57) | 0 | 0 | 0
  Leukocytes: Below (baseline) - below (Day 57) | 0 | 0 | 0
  Leukocytes: Within (baseline) - below (Day 57) | 0 | 0 | 0
  Leukocytes: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Leukocytes: Below (baseline) - within (Day 57) | 0 | 0 | 0
  Leukocytes: Within (baseline) - within (Day 57) | 20 | 22 | 21
  Leukocytes: Above (baseline) - within (Day 57) | 1 | 1 | 0
  Leukocytes: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Leukocytes: Within (baseline) - above (Day 57) | 0 | 0 | 0
  Leukocytes: Above (baseline) - above (Day 57) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - below (Day 57) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 57) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 57) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 57) | 20 | 21 | 20
  Lymphocytes: Above (baseline) - within (Day 57) | 0 | 0 | 1
  Lymphocytes: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 57) | 0 | 2 | 0
  Lymphocytes: Above (baseline) - above (Day 57) | 1 | 0 | 0
  Monocytes: Below (baseline) - below (Day 57) | 1 | 1 | 4
  Monocytes: Within (baseline) - below (Day 57) | 3 | 1 | 6
  Monocytes: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 57) | 4 | 6 | 3
  Monocytes: Within (baseline) - within (Day 57) | 13 | 15 | 8
  Monocytes: Above (baseline) - within (Day 57) | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 57) | 0 | 0 | 0
  Monocytes: Above (baseline) - above (Day 57) | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 57) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 57) | 0 | 1 | 0
  Neutrophils: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 57) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 57) | 21 | 22 | 21
  Neutrophils: Above (baseline) - within (Day 57) | 0 | 0 | 0
  Neutrophils: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 57) | 0 | 0 | 0
  Neutrophils: Above (baseline) - above (Day 57) | 0 | 0 | 0
  Platelets: Below (baseline) - below (Day 57) | 0 | 1 | 0
  Platelets: Within (baseline) - below (Day 57) | 2 | 1 | 6
  Platelets: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 57) | 0 | 1 | 0
  Platelets: Within (baseline) - within (Day 57) | 18 | 19 | 15
  Platelets: Above (baseline) - within (Day 57) | 1 | 0 | 0
  Platelets: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 57) | 0 | 1 | 0
  Platelets: Above (baseline) - above (Day 57) | 0 | 0 | 0
  ALT: Below (baseline) - below (Day 57) | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 57) | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 57) | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 57) | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 57) | 21 | 23 | 21
  ALT: Above (baseline) - within (Day 57) | 0 | 0 | 0
  ALT: Below (baseline) - above (Day 57) | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 57) | 0 | 0 | 0
  ALT: Above (baseline) - above (Day 57) | 0 | 0 | 0
  ALP: Below (baseline) - below (Day 57) | 0 | 0 | 0
  ALP: Within (baseline) - below (Day 57) | 0 | 0 | 0
  ALP: Above (baseline) - below (Day 57) | 0 | 0 | 0
  ALP: Below (baseline) - within (Day 57) | 0 | 0 | 0
  ALP: Within (baseline) - within (Day 57) | 21 | 22 | 20
  ALP: Above (baseline) - within (Day 57) | 0 | 0 | 0
  ALP: Below (baseline) - above (Day 57) | 0 | 0 | 0
  ALP: Within (baseline) - above (Day 57) | 0 | 0 | 0
  ALP: Above (baseline) - above (Day 57) | 0 | 1 | 1
  AST: Below (baseline) - below (Day 57) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 57) | 0 | 0 | 0
  AST: Above (baseline) - below (Day 57) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 57) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 57) | 20 | 20 | 20
  AST: Above (baseline) - within (Day 57) | 0 | 1 | 0
  AST: Below (baseline) - above (Day 57) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 57) | 1 | 1 | 1
  AST: Above (baseline) - above (Day 57) | 0 | 1 | 0
  BILI: Below (baseline) - below (Day 57) | 0 | 0 | 0
  BILI: Within (baseline) - below (Day 57) | 1 | 0 | 0
  BILI: Above (baseline) - below (Day 57) | 0 | 0 | 0
  BILI: Below (baseline) - within (Day 57) | 2 | 1 | 1
  BILI: Within (baseline) - within (Day 57) | 17 | 20 | 20
  BILI: Above (baseline) - within (Day 57) | 0 | 1 | 0
  BILI: Below (baseline) - above (Day 57) | 0 | 0 | 0
  BILI: Within (baseline) - above (Day 57) | 1 | 1 | 0
  BILI: Above (baseline) - above (Day 57) | 0 | 0 | 0
  BUN: Below (baseline) - below (Day 57) | 0 | 0 | 0
  BUN: Within (baseline) - below (Day 57) | 0 | 0 | 1
  BUN: Above (baseline) - below (Day 57) | 0 | 0 | 0
  BUN: Below (baseline) - within (Day 57) | 1 | 1 | 1
  BUN: Within (baseline) - within (Day 57) | 20 | 22 | 19
  BUN: Above (baseline) - within (Day 57) | 0 | 0 | 0
  BUN: Below (baseline) - above (Day 57) | 0 | 0 | 0
  BUN: Within (baseline) - above (Day 57) | 0 | 0 | 0
  BUN: Above (baseline) - above (Day 57) | 0 | 0 | 0
  CREAT: Below (baseline) - below (Day 57) | 0 | 0 | 0
  CREAT: Within (baseline) - below (Day 57) | 0 | 0 | 0
  CREAT: Above (baseline) - below (Day 57) | 0 | 0 | 0
  CREAT: Below (baseline) - within (Day 57) | 0 | 0 | 0
  CREAT: Within (baseline) - within (Day 57) | 18 | 19 | 19
  CREAT: Above (baseline) - within (Day 57) | 0 | 1 | 1
  CREAT: Below (baseline) - above (Day 57) | 0 | 0 | 0
  CREAT: Within (baseline) - above (Day 57) | 2 | 3 | 1
  CREAT: Above (baseline) - above (Day 57) | 1 | 0 | 0
  GGT: Below (baseline) - below (Day 57) | 0 | 0 | 0
  GGT: Within (baseline) - below (Day 57) | 0 | 0 | 0
  GGT: Above (baseline) - below (Day 57) | 0 | 0 | 0
  GGT: Below (baseline) - within (Day 57) | 0 | 0 | 0
  GGT: Within (baseline) - within (Day 57) | 19 | 19 | 16
  GGT: Above (baseline) - within (Day 57) | 0 | 1 | 1
  GGT: Below (baseline) - above (Day 57) | 0 | 0 | 0
  GGT: Within (baseline) - above (Day 57) | 1 | 2 | 3
  GGT: Above (baseline) - above (Day 57) | 1 | 1 | 1
  GLUC: Below (baseline) - below (Day 57) | 0 | 0 | 0
  GLUC: Within (baseline) - below (Day 57) | 0 | 0 | 0
  GLUC: Above (baseline) - below (Day 57) | 0 | 0 | 0
  GLUC: Below (baseline) - within (Day 57) | 0 | 0 | 0
  GLUC: Within (baseline) - within (Day 57) | 18 | 22 | 19
  GLUC: Above (baseline) - within (Day 57) | 0 | 0 | 0
  GLUC: Below (baseline) - above (Day 57) | 0 | 0 | 0
  GLUC: Within (baseline) - above (Day 57) | 3 | 1 | 2
  GLUC: Above (baseline) - above (Day 57) | 0 | 0 | 0
  LDH: Below (baseline) - below (Day 57) | 0 | 0 | 0
  LDH: Within (baseline) - below (Day 57) | 0 | 1 | 4
  LDH: Above (baseline) - below (Day 57) | 0 | 0 | 0
  LDH: Below (baseline) - within (Day 57) | 0 | 0 | 0
  LDH: Within (baseline) - within (Day 57) | 20 | 21 | 16
  LDH: Above (baseline) - within (Day 57) | 0 | 0 | 0
  LDH: Below (baseline) - above (Day 57) | 0 | 0 | 0
  LDH: Within (baseline) - above (Day 57) | 1 | 1 | 1
  LDH: Above (baseline) - above (Day 57) | 0 | 0 | 0
  K: Below (baseline) - below (Day 57) | 0 | 0 | 0
  K: Within (baseline) - below (Day 57) | 0 | 0 | 0
  K: Above (baseline) - below (Day 57) | 0 | 0 | 0
  K: Below (baseline) - within (Day 57) | 0 | 0 | 0
  K: Within (baseline) - within (Day 57) | 15 | 12 | 17
  K: Above (baseline) - within (Day 57) | 3 | 3 | 2
  K: Below (baseline) - above (Day 57) | 0 | 0 | 0
  K: Within (baseline) - above (Day 57) | 3 | 7 | 2
  K: Above (baseline) - above (Day 57) | 0 | 1 | 0
  Na: Below (baseline) - below (Day 57) | 0 | 0 | 0
  Na: Within (baseline) - below (Day 57) | 4 | 2 | 4
  Na: Above (baseline) - below (Day 57) | 0 | 0 | 0
  Na: Below (baseline) - within (Day 57) | 0 | 1 | 0
  Na: Within (baseline) - within (Day 57) | 17 | 20 | 17
  Na: Above (baseline) - within (Day 57) | 0 | 0 | 0
  Na: Below (baseline) - above (Day 57) | 0 | 0 | 0
  Na: Within (baseline) - above (Day 57) | 0 | 0 | 0
  Na: Above (baseline) - above (Day 57) | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Reported Reactive Arthritis or Neutropenia (AESIs)
Description: Reactive arthritis is defined as non-purulent joint inflammation that develops in response to an infection in another part of the body. Since the inflammation is triggered by a previous condition, it is termed "reactive". Intestinal pathogens that have been associated with reactive arthritis include Campylobacter, Salmonella, Yersinia, Clostridium difficile, and Shigella. If reactive arthritis is caused by an auto immune response, there is at least a possibility that it could be initiated by vaccination of susceptible people with the 1790GAHB vaccine.
Time Frame: Throughout the whole study period (from Day 1 up to Day 57)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 24
Participants
  Reactive Arthritis | 0 | 0 | 0
  Neutropenia | 2 | 3 | 1

9. Secondary Outcome: Anti-LPS S.Sonnei IgG ELISA Geometric Mean Concentrations (GMCs), by Baseline Titer
Description: Anti-LPS S.Sonnei IgG ELISA concentrations were tabulated as unadjusted geometric mean concentrations (GMCs) and expressed as ELISA units (EU) per milliliter (mL), presented with their 95% confidence intervals (CIs). Since all subjects in the study were from an endemic country, they had pre-vaccination titers equal to or above (≥) LLOQ (limit of detection).
Time Frame: At Day 1, Day 29 (28 days after the first vaccination) and Day 57 (28 days after the second vaccination)
Population: This analysis was performed on the Full Analysis Set, including subjects with at least 1 dose of study vaccine administered. Numbers decreased over time, hence at study Visit 5 (Day 57), not all subjects from study Visit 1 (Day 1) had available immunogenicity results.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 24
EU/mL
  Day 1 | 971 [519 to 1817] | 1196 [750 to 1909] | 994 [547 to 1809]
  Day 29: number analyzed (Participants) | 22 | 26 | 22
  Day 29 | 2038 [1324 to 3135] | 5301 [3598 to 7810] | 1100 [572 to 2115]
  Day 57: number analyzed (Participants) | 21 | 23 | 21
  Day 57 | 3030 [1909 to 4809] | 4706 [3391 to 6531] | 987 [507 to 1922]

10. Secondary Outcome: Anti-LPS S. Sonnei Geometric Mean Ratios (GMRs) Between Post- and Pre-vaccination Samples
Description: The ratio was expressed as unadjusted geometric mean ratio (GMR) and presented with its 95% confidence interval (CI).
Time Frame: At Day 1, Day 29 (28 days after the first vaccination) and Day 57 (28 days after the second vaccination)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 22
Geometric mean ratio
  At Day 29 versus Day 1 | 2.1 [1.31 to 3.36] | 4.43 [2.94 to 6.67] | 1.06 [0.91 to 1.24]
  At Day 57 versus Day 1: number analyzed (Participants) | 21 | 23 | 21
  At Day 57 versus Day 1 | 3.1 [2.29 to 4.2] | 4.3 [3.02 to 6.12] | 1.07 [0.91 to 1.25]
  At Day 57 versus Day 29: number analyzed (Participants) | 21 | 23 | 21
  At Day 57 versus Day 29 | 1.44 [1.09 to 1.89] | 1.02 [0.9 to 1.16] | 1.01 [0.8 to 1.26]

11. Secondary Outcome: Number of Subjects With Seroresponse to Anti-LPS S. Sonnei IgG ELISA, by Baseline Titer
Description: Seroresponse was defined as: if the baseline value was greater than 50 EU then an increase of at least 50% in the post-vaccination sample as compared to baseline (i.e., [{post-vac minus baseline}/baseline]100% ≥ 50%); if the baseline value was less or equal to 50 EU then an increase of at least 25 EU in the post-vaccination sample as compared to baseline (i.e., [post-vac minus baseline] ≥ 25 EU).
  Since all subjects in the study were from an endemic country, they had pre-vaccination titers equal to or above (≥) LLOQ (limit of detection).
Time Frame: At Day 29 (28 days after the first vaccination) and Day 57 (28 days after the second vaccination)
Population: This analysis was based on the Full Analysis Set, including subjects with at least 1 dose of study vaccine administered. Some subjects were excluded due to implausible values from all study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 22
Participants
  Anti-LPS, Day 29 | 15 | 25 | 2
  Anti-LPS, Day 57: number analyzed (Participants) | 21 | 23 | 21
  Anti-LPS, Day 57 | 19 | 22 | 1

12. Secondary Outcome: Number of Subjects With Titers Post Vaccination Concentration for Anti-LPS S. Sonnei ≥ 121 U/mL
Description: The analysis cut-off value (121 U/mL) was expressed in units per milliliter (U/mL), as assessed by the Enzyme-Linked Immunosorbent Assay (ELISA).
Time Frame: At Day 1, Day 29 (28 days after the first vaccination) and Day 57 (28 days after the second vaccination)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
Number analyzed (Participants) | 22 | 26 | 22
Participants
  Day 1 | 21 | 24 | 21
  Day 29 | 22 | 26 | 19
  Day 57: number analyzed (Participants) | 21 | 23 | 21
  Day 57 | 21 | 23 | 19

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during 7 days following each vaccination; Unsolicited AEs: during 28 days following each vaccination; SAEs: throughout the whole study period (from Day 1 up to Day 57).
Arm/Group | 1790GAHB 25 μg Group | 1790GAHB 100 μg Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/22 | 3/26 | 1/24
Other Adverse Events (participants affected / at risk) | 22/22 | 26/26 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1790GAHB 25 μg Group (N=22) | 1790GAHB 100 μg Group (N=26) | Control Group (N=24)
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 1 — Neutropenia was considered as an AE of specific interest and for reporting purpose systematically reported as an SAE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1790GAHB 25 μg Group (N=22) | 1790GAHB 100 μg Group (N=26) | Control Group (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chills (General disorders) | 5 | 5 | 5
Fatigue (General disorders) | 3 | 9 | 9
Induration (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 21 | 25 | 19
Malaise (General disorders) | 3 | 3 | 10
Pyrexia (General disorders) | 1 | 1 | 1
Bone tuberculosis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 2
Furuncle (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Genital herpes (Infections and infestations) | 1 | 0 | 0
Malaria (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 2
Pyuria (Infections and infestations) | 1 | 0 | 2
Rhinitis (Infections and infestations) | 1 | 1 | 2
Sinusitis (Infections and infestations) | 3 | 3 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 1
Urinary tract infection (Infections and infestations) | 1 | 4 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 5
Limb discomfort (Musculoskeletal and connective tissue disorders) | 5 | 7 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 7
Dizziness (Nervous system disorders) | 1 | 2 | 2
Headache (Nervous system disorders) | 11 | 14 | 11
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 15 | 18 | 14
Injection site induration (General disorders) | 17 | 22 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT02676895/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT02676895/SAP_001.pdf